CLINICAL TRIAL: NCT02596945
Title: Non-Interventional Observation Trial to Investigate the Efficacy, Safety and Usability of Mircera in PD Patients in Daily Use
Brief Title: Observational Study of Methoxy Polyethylene Glycol Epoetin Beta Daily Use in Participants on Peritoneal Dialysis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22000
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-05

CONDITIONS: Renal Impairment; Renal Anemia of Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Peritoneal Dialysis participants: Participants who are on peritoneal dialysis and have been prescribed with methoxy polyethylene glycol were observed for a period of 9 months.
  Interventions: Drug: Methoxy polyethylene glycol epoetin beta

INTERVENTIONS:
Drug: Methoxy polyethylene glycol epoetin beta — Methoxy polyethylene glycol epoetin beta is prescribed as per physician's discretion in accordance with the Summary of Product Characteristics (SmPC).
  Other Names: Mircera

SUMMARY:
This non-interventional, observational study investigates the efficacy, safety and usability of methoxy polyethylene glycol epoetin beta in participants on peritoneal dialysis. Participants who were prescribed methoxy polyethylene glycol epoetin beta by their doctor and who meet the selection criteria were to be enrolled and documented in this study for a period of 9 months of treatment with methoxy polyethylene glycol epoetin beta with respect to efficacy, safety and usability.

ELIGIBILITY:
Inclusion Criteria:

* Participants on peritoneal dialysis
* Need for Erythropoiesis Stimulating Agent (ESA) therapy
* Prescription of methoxy polyethylene glycol epoetin beta by the doctor

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants on peritoneal dialysis who are in need of ESA therapy and have been prescribed methoxy polyethylene glycol beta by the doctor
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2009-07-31 (Actual); Primary Completion 2011-02-28 (Actual); Study Completion 2011-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Dres. Michael Koch Hannelore Klimke Wolfgang Kulas u.w., Mettmann, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Peritoneal Dialysis Participants: Participants who were on peritoneal dialysis and prescribed methoxy polyethylene glycol epoetin beta as per physician's discretion in accordance with the Summary of Product Characteristics (SmPC) were observed for a period of 9 months.
Period: Overall Study
Arm/Group | Peritoneal Dialysis Participants
Started | 223
Treated | 220
Completed | 167
Not Completed | 56
Not completed — No documentation of study drug dosing | 3
Not completed — Other | 32
Not completed — Change to hemodialysis | 15
Not completed — Other Erythropoietin stimulating agent | 4
Not completed — Withdrawal by Subject | 1
Not completed — Missing | 1

BASELINE CHARACTERISTICS:
Population: Safety Set (SS) population: Participants who received at least 1 dose of study drug were included.
Groups:
- Peritoneal Dialysis Participants: Participants who were on peritoneal dialysis and prescribed methoxy polyethylene glycol epoetin beta as per physician's discretion in accordance with the SmPC were observed for a period of 9 months.
Arm/Group | Peritoneal Dialysis Participants
Number analyzed (Participants) | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107
  Male | 113

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hemoglobin Values in the Range of 11-12 Grams Per Deciliter (g/dL) During the Evaluation Period of Visit 7 (Month 7) to Visit 9 (Month 9)
Time Frame: Month 7 to Month 9
Population: Modified Efficacy Set (MES) population (All participants who received at least 1 dose of study drug and for whom at least 2 hemoglobin measurements were available during the evaluation period (Month 7 to Month 9).
Measure: Number; unit: percentage of participants
Arm/Group | Peritoneal Dialysis Participants
Number analyzed (Participants) | 162
percentage of participants | 14.8

2. Secondary Outcome: Percentage of Participants With Hemoglobin Values in the Range of 11-13 g/dL During the Evaluation Period of Visit 7 (Month 7) to Visit 9 (Month 9)
Time Frame: Month 7 to Month 9
Population: MES population.
Measure: Number; unit: percentage of participants
Arm/Group | Peritoneal Dialysis Participants
Number analyzed (Participants) | 162
percentage of participants | 38.9

3. Secondary Outcome: Average Duration in Days Mircera Was Administered at a Stable Dose
Time Frame: Up to 9 months
Population: MES population.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Peritoneal Dialysis Participants
Number analyzed (Participants) | 162
days | 182.1 (122.7)

ADVERSE EVENTS:
Time Frame: Up to 20 months
Description: Only adverse drug reactions (ADRs) were planned to be reported per protocol for this study and since there were no ADR observed, adverse events were also not observed.
Arm/Group | Peritoneal Dialysis Participants
Serious Adverse Events (participants affected / at risk) | 0/220
Other Adverse Events (participants affected / at risk) | 0/220

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.